CLINICAL TRIAL: NCT03366428
Title: Phase 1, Multicenter, Open-label, Multiple-dose Study of DS-8201a to Assess the Effect on the QT Interval and Pharmacokinetics in Subjects With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Brief Title: Phase 1 Study to Evaluate the Effect of DS-8201a on the QT/QTc Interval and Pharmacokinetics in HER2-Expressing Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-J102; 173791 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Malignant Neoplasm of Breast
Keywords: HER2; Breast cancer; Oncology; Antibody drug conjugate; ADC
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All participants will receive DS-8201a by intravenous infusion
  Interventions: Drug: DS-8201a

INTERVENTIONS:
Drug: DS-8201a — DS-8201a is supplied as a lyophilized powder which is reconstituted for infusion
  Other Names: Experimental product

SUMMARY:
This study will look at the effect on the QTc interval and pharmacokinetics after multiple dosing in subjects with HER2-expressing metastatic and/or unresectable breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has a pathologically documented unresectable or metastatic breast cancer with HER2 expression (immunohistochemistry [IHC] 3+, IHC 2+, IHC 1+ and/or in situ hybridization [ISH] +) that is refractory to or intolerable with standard treatment, or for which no standard treatment is available
* Has a left ventricular ejection fraction (LVEF) ≥ 50%
* Has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1

Exclusion Criteria:

* Has a medical history of myocardial infarction within 6 months before enrollment
* Has a medical history of ventricular arrhythmias, other than rare occasional premature ventricular contractions
* Has uncontrolled or significant cardiovascular disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (7):
- Japan (7):
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Koto-Ku, Tokyo
  - Toranomon Hospital, Minato-Ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Social Medical Corporation Hakuaikai Sagara Hospital, Kagoshima
  - Shizuoka Cancer Center, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Shimomura A, Takano T, Takahashi S, Sagara Y, Watanabe J, Tokunaga E, Shinkai T, Kamio T, Kikumori K, Kamiyama E, Fujisaki Y, Saotome D, Yamashita T. Effect of Trastuzumab Deruxtecan on QT/QTc Interval and Pharmacokinetics in HER2-Positive or HER2-Low Metastatic/Unresectable Breast Cancer. Clin Pharmacol Ther. 2023 Jan;113(1):160-169. doi: 10.1002/cpt.2757. Epub 2022 Oct 18. PMID 36164935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 participants who met all inclusion criteria and no exclusion criteria were enrolled and treated at 7 sites in Japan.
Pre-assignment Details: The 6.4 mg/kg DS-8201a dose was chosen for this study based on the efficacy, safety, and pharmacokinetic profiles established in an earlier Phase 1 trial.
Groups:
- DS-8201a: Participants who received 6.4 mg/kg of DS-8201a as an intravenous (IV) infusion once every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | DS-8201a
Started | 51
Completed | 0
Not Completed | 51
Not completed — Progressive disease per RECIST v1.1 | 33
Not completed — Adverse Event | 12
Not completed — Clinical progression | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- DS-8201a: Participants who received 6.4 mg/kg of DS-8201a as an intravenous (IV) infusion once every 3 weeks on Day 1 of each 21-day cycle.
Arm/Group | DS-8201a
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.48)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 38
  ≥65 | 13
  >75 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 51
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 51

OUTCOME MEASURES:

1. Primary Outcome: Changes in QTcF After Treatment With DS-8201a in Participants With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Description: The number of participants with notable electrocardiogram changes meeting predefined criteria is being reported.
Time Frame: Screening (within 7 days before enrollment) up to Cycle 3 Day 15 (each cycle is 21 days)
Population: QTc and QTcF were assessed in the Cardiac Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a
Number analyzed (Participants) | 49
Participants
  Maximum change from baseline in QTcF: >30 ms | 3
  Maximum change from baseline in QTcF: >60 ms | 0

2. Primary Outcome: Pharmacokinetic Parameters of Maximum Serum Concentration (Cmax) After Cycle 1 and Cycle 3 Treatments With DS-8201a in Participants With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Description: Maximum serum concentration (Cmax) of DS-8201a and total anti-HER2 antibody was assessed.
Time Frame: Cycles 1 and 3: Day 1: before infusion (BI), end of infusion (EOI), 2 hours, 4 hours, 7 hours; Days 2 and 4: 24 hours, 72 hours; Days 8 and 15; Cycle 2: Day 1 BI, EOI; Cycles 4, 6, and 8: Day 1 BI and EOI (each cycle is 21 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | DS-8201a
Number analyzed (Participants) | 51
ug/mL
  DS-8201: Cycle 1 | 179 (112)
  DS-8201: Cycle 3: number analyzed (Participants) | 37
  DS-8201: Cycle 3 | 154 (23.3)
  Total Anti-HER2 antibody: Cycle 1 | 165 (110)
  Total Anti-HER2 antibody: Cycle 3: number analyzed (Participants) | 37
  Total Anti-HER2 antibody: Cycle 3 | 142 (27.0)

3. Primary Outcome: Pharmacokinetic Parameters of Maximum Serum Concentration (Cmax) of MAAA-1181 After Cycle 1 and Cycle 3 Treatments With DS-8201a in Participants With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Description: Maximum serum concentration (Cmax) of MAAA-1181 was assessed.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-8201a
Number analyzed (Participants) | 51
ng/mL
  MAAA-1181a: Cycle 1 | 12.6 (4.49)
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 37
  MAAA-1181a: Cycle 3 | 9.60 (3.89)

4. Primary Outcome: Pharmacokinetic Parameters Area Under the Concentration-Time Curve After Cycle 1 and Cycle 3 Treatments With DS-8201a in Participants With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Description: Area under the concentration versus-time curve from time 0 to the last quantifiable concentration (AUClast) and during the dosing interval (AUCtau) of DS-8201a and total anti-HER2 antibody were assessed.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | DS-8201a
Number analyzed (Participants) | 51
ug*d/mL
  AUClast, DS-8201: Cycle 1 | 677 (143)
  AUClast, Total Anti-HER2 antibody: Cycle 1 | 753 (190)
  AUCtau, DS-8201: Cycle 1 | 677 (141)
  AUCtau, DS-8201: Cycle 3: number analyzed (Participants) | 37
  AUCtau, DS-8201: Cycle 3 | 905 (189)
  AUCtau, Total Anti-HER2 antibody: Cycle 1 | 752 (185)
  AUCtau, Total Anti-HER2 antibody: Cycle 3: number analyzed (Participants) | 37
  AUCtau, Total Anti-HER2 antibody: Cycle 3 | 1030 (256)

5. Primary Outcome: Pharmacokinetic Parameters Area Under the Concentration-Time Curve of MAAA-1181 After Cycle 1 and Cycle 3 Treatments With DS-8201a in Participants With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Description: Area under the concentration versus-time curve from time 0 to the last quantifiable concentration (AUClast) and during the dosing interval (AUCtau) were assessed.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | DS-8201a
Number analyzed (Participants) | 51
ng*d/mL
  AUClast, MAAA-1181a: Cycle 1 | 39.3 (11.3)
  AUCtau, MAAA-1181a: Cycle 1 | 39.0 (11.2)
  AUCtau, MAAA-1181a: Cycle 3: number analyzed (Participants) | 37
  AUCtau, MAAA-1181a: Cycle 3 | 41.5 (13.8)

6. Secondary Outcome: Objective Response Rate Based on The Investigator's Assessment (Unconfirmed) Following DS-8201a Treatment in Participants With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Description: Objective response rate (ORR) was defined as unconfirmed complete response (CR) and partial response (PR) as assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 12 months post-dose
Population: Response was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- HER2 Positive: Participants with HER2 positive expression (defined as immunohistochemistry 3+ or in situ hybridization positive) who received 6.4 mg/kg of DS-8201a as an intravenous (IV) infusion once every 3 weeks on Day 1 of each 21-day cycle.
- HER2 Low: Participants with HER2 low expression (defined as immunohistochemistry 1+ or 2+/ in situ hybridization negative or missing) who received 6.4 mg/kg of DS-8201a as an intravenous (IV) infusion once every 3 weeks on Day 1 of each 21-day cycle.
Arm/Group | HER2 Positive | HER2 Low
Number analyzed (Participants) | 4 | 47
Participants | 2 | 18

7. Secondary Outcome: Objective Response Rate Based on The Investigator's Assessment (Unconfirmed) Following DS-8201a Treatment in Participants With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Description: as for outcome 6
Time Frame: Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 38 months post-dose
Population: Response was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | HER2 Positive | HER2 Low
Number analyzed (Participants) | 4 | 47
Participants | 2 | 23

8. Secondary Outcome: Treatment-Emergent Adverse Events of Any Grade by System Organ Classes and Preferred Term Following DS-8201a Treatment in Participants With HER2-expressing Metastatic and/or Unresectable Breast Cancer
Description: Adverse events (AEs) were to be coded using MedDRA Version 20.1 and assigned severity grades based on Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. A treatment-emergent adverse event (TEAE) was defined as an AE that occurred, having been absent before the first dose of study drug, or had worsened in severity or seriousness after initiating the study drug until 47 days after last dose of study drug.
Time Frame: Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to approximately 12 months post-dose
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a
Number analyzed (Participants) | 51
Participants
  Any TEAEs | 51
  Gastrointestinal Disorders | 45
  Nausea | 42
  Vomiting | 20
  Constipation | 16
  Stomatitis | 16
  Diarrhoea | 14
  Investigations | 45
  Neutrophil count decreased | 36
  White blood cell count decreased | 31
  Platelet count decreased | 20
  Lymphocyte count decreased | 13
  Alanine aminotransferase increased | 12
  Aspartate aminotransferase increased | 12
  Blood and Lymphatic System Disorders | 30
  Anaemia | 30
  Skin and Subcutaneous Tissue Disorders | 27
  Alopecia | 21
  General Disorders and Administration Site Conditions | 25
  Fatigue | 11
  Infections and Infestations | 21
  Nasopharyngitis | 11
  Metabolism and Nutrition Disorders | 19
  Decreased appetite | 16
  Nervous System Disorders | 15
  Respiratory, Thoracic, and Mediastinal Disorders | 12

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 38 months post-dose.
Arm/Group | DS-8201a
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 9/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8201a (N=51)
Nausea (Gastrointestinal disorders) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Cellulitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8201a (N=51)
Nausea (Gastrointestinal disorders) | 42
Neutrophil count decreased (Investigations) | 36
White blood cell count decreased (Investigations) | 34
Anaemia (Blood and lymphatic system disorders) | 32
Alopecia (Skin and subcutaneous tissue disorders) | 21
Platelet count decreased (Investigations) | 20
Vomiting (Gastrointestinal disorders) | 21
Constipation (Gastrointestinal disorders) | 17
Stomatitis (Gastrointestinal disorders) | 21
Decreased appetite (Metabolism and nutrition disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 17
Lymphocyte count decreased (Investigations) | 15
Alanine aminotransferase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 13
Fatigue (General disorders) | 11
Nasopharyngitis (Infections and infestations) | 16
Malaise (General disorders) | 12
Pyrexia (General disorders) | 14
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Electrocardiogram QT prolonged (Investigations) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Anxiety (Psychiatric disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5
Insomnia (Psychiatric disorders) | 5
Weight decreased (Investigations) | 5
Lung infection (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 5
Ginsivitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Paronychia (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Angular cheilitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Dacryocystitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Skin candida (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seasonal allergy (Immune system disorders) | 2
Allergy to arthropod sting (Immune system disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Agitation (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 2
Akathisia (Nervous system disorders) | 1
Vagus nerve disorder (Nervous system disorders) | 1
Visual perseveration (Nervous system disorders) | 1
Conjunctivitis allergic (Eye disorders) | 2
Dry eye (Eye disorders) | 2
Punctate keratitis (Eye disorders) | 2
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Corneal disorder (Eye disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Palpitations (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 3
Proctalgia (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2
Faeces soft (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 3
Chest pain (General disorders) | 2
Withdrawal syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Blood alkaline phosphatase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 4
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Protein total decreased (Investigations) | 2
Blood urea increased (Investigations) | 1
Weight increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Bite (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03366428/Prot_SAP_000.pdf